CLINICAL TRIAL: NCT03443050
Title: Training on Unstable Surfaces and Effects on the Balance of Healthy Young People, a Randomized Clinical Trial
Brief Title: Training on Unstable Surfaces and Effects on the Balance of Healthy Young People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Jose María Blasco Igual, Principal Investigator, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: UNSTABLE_UV
Record Dates: First submitted 2018-02-07; First posted 2018-02-22 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Balance training on unstable surfaces
  Interventions: Other: Unstable
- Control (Active Comparator): Balance training on stable surface
  Interventions: Other: Stable

INTERVENTIONS:
Other: Unstable — This group will train over unstable surfaces to enhance balance abilities
  Other Names: Experimental
  Arms: Experimental
Other: Stable — This group will train over stable surface to enhance balance abilities
  Other Names: Control
  Arms: Control

SUMMARY:
The objective of this study is to determine the effects on balance and postural control produced by the implementation of a training program that includes work with unstable surfaces in its methods. It also seeks to quantify to what extent the benefits exceed those achieved with a training of similar characteristics, but implemented on a stable surface. An intensive program is proposed, whose target population is young adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy young adults aged between 18 and 30

Exclusion Criteria:

* Professional athlete
* Musculoskeletal injury in the last 12 months (i.e. sprain, bone fracture)
* Known balance disorders including vertigo, central or vestibular limitations

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-04-04 (Actual); Study Completion 2018-04-04 (Actual)

PRIMARY OUTCOMES:
Y-balance test | change from baseline to end of intervention (4weeks)
  Dynamic balance. The maximum length in cm achieved for each leg in the anterior, posterior-lateral and medial-lateral positions will be recorded.

SECONDARY OUTCOMES:
Posturography (1) | change from baseline to end of intervention (4weeks)
  A force T-plate platform will be used to assess posture in terms of sway area (mm2)
Posturography (2) | change from baseline to end of intervention (4weeks)
  A force T-plate platform will be used to assess posture in terms of mean velocity (m/s)
Emery test | change from baseline to end of intervention (4weeks)
  Static balance and proprioception as measured with the eyes closed to keep balance with one leg over an Airex(R) balance pad. The time in seconds will be recorded.
Functional reach | change from baseline to end of intervention (4weeks)
  Test of stability, measured as the distance reached when leaning forward without falling (cm)

OTHER OUTCOMES:
Jumping sideways test | change from baseline to end of intervention (4weeks)
  Test of agility. Evaluates motor coordination under the pressure of time of implementation. The jumps in 15 seconds are recorded
T-agility test | change from baseline to end of intervention (4weeks)
  Evaluation of the performance of the change of direction, as well as the speed and power of the lower extremities

CONTACTS AND LOCATIONS:
Overall Officials: Jose M Blasco, PhD, Principal Investigator — University of Valencia
Locations (1):
- University of Valencia. Facultat de Fisioterapia, Valencia, Spain